CLINICAL TRIAL: NCT03876054
Title: Long-Term Real-World Outcomes Study on Patients Implanted With a Neurostimulator
Acronym: REALITY
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10279
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
Keywords: spinal cord stimulation; dorsal root ganglion stimulation
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Spinal cord stimulation (SCS): Subjects using Abbott SCS systems
  Interventions: Device: Spinal cord stimulation (SCS)
- Dorsal root ganglion stimulation (DRG): Subjects using Abbott DRG system
  Interventions: Device: Dorsal root ganglion stimulation (DRG)

INTERVENTIONS:
Device: Spinal cord stimulation (SCS) — Subjects will be implanted with market-released Abbott SCS systems
  Groups: Spinal cord stimulation (SCS)
Device: Dorsal root ganglion stimulation (DRG) — Subjects will be implanted with market-released Abbott DRG system
  Groups: Dorsal root ganglion stimulation (DRG)

SUMMARY:
The REALITY study is a prospective, post-market, non-randomized, multi-center, single-arm, open-label study intended to collect short- and long-term safety and effectiveness data on various populations implanted with Abbott's neurostimulation systems.

DETAILED DESCRIPTION:
This study has broad inclusion criteria and minimal exclusion criteria to ensure the results are representative of the real-world use of these devices. Enrollment caps will be implemented to ensure patients from approved indications are represented. Individuals who are scheduled to receive an implantable Abbott neurostimulation system are eligible for study consideration. The study will enroll up to 2,000 subjects from up to 100 participating centers. Subject enrollment is expected to be completed within 7 years; subjects will be followed for 5 years. The total duration of the study is expected to be 13 years, including enrollment, data collection from all subjects, and study close out.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to any clinical investigation related procedure.
2. Subject is at least 18 years (or the minimum age required by local law to consent for participation in a clinical investigation) or older at the time of enrollment.
3. Subject is scheduled to have an Abbott neurostimulation system implanted within 60 days of baseline.
4. Subject has a baseline (with no stimulation) pain NRS of ≥ 6.

Exclusion Criteria:

1. Subject is enrolled, or intends to participate, in a competing clinical study, as determined by Abbott.
2. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements.
3. Subject has or is scheduled to receive an intrathecal pump.
4. Subject is part of a vulnerable population.
5. Subject has an existing implanted neuromodulation device to address their chronic pain.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This clinical investigation will enroll adult male and female individuals scheduled to have an Abbott neurostimulation system implanted. Subjects must meet all eligibility criteria and provide written informed consent prior to conducting any investigation-specific procedures not considered standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Rate of device and procedure related adverse events, deaths, and device deficiencies | Baseline
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | Permanent Implant Procedure
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | 6 months
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | 9 months
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be assessed via Telephone Calls and will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | 1 Year
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | 1.5 Years
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be assessed via Telephone Calls and will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | 2 Years
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | 2.5 Years
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be assessed via Telephone Calls and will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | 3 Years
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | 3.5 Years
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be assessed via Telephone Calls and will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | 4 Years
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | 4.5 Years
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be assessed via Telephone Calls and will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of device and procedure related adverse events, deaths, and device deficiencies | 5 Years
  Serious adverse device effects (SADEs), adverse device effects (ADEs), deaths, and device deficiencies will be summarized using counts, percentages or Kaplan-Meier survival estimates.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.

OTHER OUTCOMES:
Mean Change in Clinical improvement from baseline to each follow up visit assessed by PROMIS-29 | 6 months
  The PROMIS-29 is used to estimate overall quality of life by assessing the following domains known to impact activities of daily living: physical function, sleep disturbance, depression, anxiety, fatigue, pain interference, pain intensity, and social role satisfaction. The scale requires subjects to rate the frequency and/or severity of symptoms and experiences related to each of these domains. The final item is an 11-point pain intensity numerical rating scale (NRS) by which the subject rates their average pain over the past 7 days. Subjects should read each item and check the one box that most closely represents their response.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by PROMIS-29 | 1 Year
  The PROMIS-29 is used to estimate overall quality of life by assessing the following domains known to impact activities of daily living: physical function, sleep disturbance, depression, anxiety, fatigue, pain interference, pain intensity, and social role satisfaction. The scale requires subjects to rate the frequency and/or severity of symptoms and experiences related to each of these domains. The final item is an 11-point pain intensity numerical rating scale (NRS) by which the subject rates their average pain over the past 7 days. Subjects should read each item and check the one box that most closely represents their response.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by PROMIS-29 | 2 Years
  The PROMIS-29 is used to estimate overall quality of life by assessing the following domains known to impact activities of daily living: physical function, sleep disturbance, depression, anxiety, fatigue, pain interference, pain intensity, and social role satisfaction. The scale requires subjects to rate the frequency and/or severity of symptoms and experiences related to each of these domains. The final item is an 11-point pain intensity numerical rating scale (NRS) by which the subject rates their average pain over the past 7 days. Subjects should read each item and check the one box that most closely represents their response.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by PROMIS-29 | 3 Years
  The PROMIS-29 is used to estimate overall quality of life by assessing the following domains known to impact activities of daily living: physical function, sleep disturbance, depression, anxiety, fatigue, pain interference, pain intensity, and social role satisfaction. The scale requires subjects to rate the frequency and/or severity of symptoms and experiences related to each of these domains. The final item is an 11-point pain intensity numerical rating scale (NRS) by which the subject rates their average pain over the past 7 days. Subjects should read each item and check the one box that most closely represents their response.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by PROMIS-29 | 4 Years
  The PROMIS-29 is used to estimate overall quality of life by assessing the following domains known to impact activities of daily living: physical function, sleep disturbance, depression, anxiety, fatigue, pain interference, pain intensity, and social role satisfaction. The scale requires subjects to rate the frequency and/or severity of symptoms and experiences related to each of these domains. The final item is an 11-point pain intensity numerical rating scale (NRS) by which the subject rates their average pain over the past 7 days. Subjects should read each item and check the one box that most closely represents their response.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by PROMIS-29 | 5 Years
  The PROMIS-29 is used to estimate overall quality of life by assessing the following domains known to impact activities of daily living: physical function, sleep disturbance, depression, anxiety, fatigue, pain interference, pain intensity, and social role satisfaction. The scale requires subjects to rate the frequency and/or severity of symptoms and experiences related to each of these domains. The final item is an 11-point pain intensity numerical rating scale (NRS) by which the subject rates their average pain over the past 7 days. Subjects should read each item and check the one box that most closely represents their response.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Numerical Rating Score (NRS) | 6 months
  The pain NRS consists of 1 question that will be asked by interviewing the subjects. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their pain at the time of study visit specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Numerical Rating Score (NRS) | 9 months
  The pain NRS consists of 1 question that will be asked to the subjects via telephone calls. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their pain at the time of study visit specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Numerical Rating Score (NRS) | 1 year
  The pain NRS consists of 1 question that will be asked by interviewing the subjects. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their pain at the time of study visit specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Numerical Rating Score (NRS) | 1.5 years
  The pain NRS consists of 1 question that will be asked to the subjects via telephone calls. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their pain at the time of study visit specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Numerical Rating Score (NRS) | 2 Years
  The pain NRS consists of 1 question that will be asked by interviewing the subjects. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their pain at the time of study visit specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Numerical Rating Score (NRS) | 2.5 Years
  The pain NRS consists of 1 question that will be asked to the subjects via telephone calls. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their pain at the time of study visit specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Numerical Rating Score (NRS) | 3 Years
  The pain NRS consists of 1 question that will be asked by interviewing the subjects. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their pain at the time of study visit specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Numerical Rating Score (NRS) | 3.5 Years
  The pain NRS consists of 1 question that will be asked to the subjects via telephone calls. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their pain at the time of study visit specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Numerical Rating Score (NRS) | 4 Years
  The pain NRS consists of 1 question that will be asked by interviewing the subjects. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their pain at the time of study visit specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Numerical Rating Score (NRS) | 4.5 Years
  The pain NRS consists of 1 question that will be asked to the subjects via telephone calls. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their pain at the time of study visit specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Numerical Rating Score (NRS) | 5 Years
  The pain NRS consists of 1 question that will be asked by interviewing the subjects. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their pain at the time of study visit specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Catastrophizing Scale (PCS) | 6 months
  Pain Catastrophizing Scale is a validated scale that measures the magnitude of catastrophizing (negative thoughts and feelings while a patient is experiencing pain). Subjects answer questions about how they feel and what they think about when they are in pain (i.e., not at the current moment). The scale includes 13 statements concerning pain experiences that are rated on a scale between 0 'not at all' and 4 'all the time'. The scale is self-administered and takes 5 minutes to complete. A higher score indicates a higher level of catastrophizing.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Catastrophizing Scale (PCS) | 1 Year
  Pain Catastrophizing Scale is a validated scale that measures the magnitude of catastrophizing (negative thoughts and feelings while a patient is experiencing pain). Subjects answer questions about how they feel and what they think about when they are in pain (i.e., not at the current moment). The scale includes 13 statements concerning pain experiences that are rated on a scale between 0 'not at all' and 4 'all the time'. The scale is self-administered and takes 5 minutes to complete. A higher score indicates a higher level of catastrophizing.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Catastrophizing Scale (PCS) | 2 Years
  Pain Catastrophizing Scale is a validated scale that measures the magnitude of catastrophizing (negative thoughts and feelings while a patient is experiencing pain). Subjects answer questions about how they feel and what they think about when they are in pain (i.e., not at the current moment). The scale includes 13 statements concerning pain experiences that are rated on a scale between 0 'not at all' and 4 'all the time'. The scale is self-administered and takes 5 minutes to complete. A higher score indicates a higher level of catastrophizing.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Catastrophizing Scale (PCS) | 3 Years
  Pain Catastrophizing Scale is a validated scale that measures the magnitude of catastrophizing (negative thoughts and feelings while a patient is experiencing pain). Subjects answer questions about how they feel and what they think about when they are in pain (i.e., not at the current moment). The scale includes 13 statements concerning pain experiences that are rated on a scale between 0 'not at all' and 4 'all the time'. The scale is self-administered and takes 5 minutes to complete. A higher score indicates a higher level of catastrophizing.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Catastrophizing Scale (PCS) | 4 Years
  Pain Catastrophizing Scale is a validated scale that measures the magnitude of catastrophizing (negative thoughts and feelings while a patient is experiencing pain). Subjects answer questions about how they feel and what they think about when they are in pain (i.e., not at the current moment). The scale includes 13 statements concerning pain experiences that are rated on a scale between 0 'not at all' and 4 'all the time'. The scale is self-administered and takes 5 minutes to complete. A higher score indicates a higher level of catastrophizing.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Pain Catastrophizing Scale (PCS) | 5 Years
  Pain Catastrophizing Scale is a validated scale that measures the magnitude of catastrophizing (negative thoughts and feelings while a patient is experiencing pain). Subjects answer questions about how they feel and what they think about when they are in pain (i.e., not at the current moment). The scale includes 13 statements concerning pain experiences that are rated on a scale between 0 'not at all' and 4 'all the time'. The scale is self-administered and takes 5 minutes to complete. A higher score indicates a higher level of catastrophizing.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Oswestry Disability Index (ODI) | 6 months
  The ODI is a 10-item scale that evaluates disability related to low-back and leg pain. It is widely used, validated, and has been translated into several languages. Each section in the scale covers a different domain (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling). Each item is scored on a scale from 0-5 with the first item scored a "0" and representing no disability. The final item is scored a "5" and represents the maximum level of disability. If more than one response in a section is checked, the highest score is chosen. The scores for each section are summed for a final score ranging from 0 to 50. If an item is not answered, the total score is instead calculated as a percentage of the total possible score for all items that were completed.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Oswestry Disability Index (ODI) | 1 Year
  The ODI is a 10-item scale that evaluates disability related to low-back and leg pain. It is widely used, validated, and has been translated into several languages. Each section in the scale covers a different domain (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling). Each item is scored on a scale from 0-5 with the first item scored a "0" and representing no disability. The final item is scored a "5" and represents the maximum level of disability. If more than one response in a section is checked, the highest score is chosen. The scores for each section are summed for a final score ranging from 0 to 50. If an item is not answered, the total score is instead calculated as a percentage of the total possible score for all items that were completed.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Oswestry Disability Index (ODI) | 2 Years
  The ODI is a 10-item scale that evaluates disability related to low-back and leg pain. It is widely used, validated, and has been translated into several languages. Each section in the scale covers a different domain (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling). Each item is scored on a scale from 0-5 with the first item scored a "0" and representing no disability. The final item is scored a "5" and represents the maximum level of disability. If more than one response in a section is checked, the highest score is chosen. The scores for each section are summed for a final score ranging from 0 to 50. If an item is not answered, the total score is instead calculated as a percentage of the total possible score for all items that were completed.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Oswestry Disability Index (ODI) | 3 Years
  The ODI is a 10-item scale that evaluates disability related to low-back and leg pain. It is widely used, validated, and has been translated into several languages. Each section in the scale covers a different domain (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling). Each item is scored on a scale from 0-5 with the first item scored a "0" and representing no disability. The final item is scored a "5" and represents the maximum level of disability. If more than one response in a section is checked, the highest score is chosen. The scores for each section are summed for a final score ranging from 0 to 50. If an item is not answered, the total score is instead calculated as a percentage of the total possible score for all items that were completed.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Oswestry Disability Index (ODI) | 4 Years
  The ODI is a 10-item scale that evaluates disability related to low-back and leg pain. It is widely used, validated, and has been translated into several languages. Each section in the scale covers a different domain (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling). Each item is scored on a scale from 0-5 with the first item scored a "0" and representing no disability. The final item is scored a "5" and represents the maximum level of disability. If more than one response in a section is checked, the highest score is chosen. The scores for each section are summed for a final score ranging from 0 to 50. If an item is not answered, the total score is instead calculated as a percentage of the total possible score for all items that were completed.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Oswestry Disability Index (ODI) | 5 Years
  The ODI is a 10-item scale that evaluates disability related to low-back and leg pain. It is widely used, validated, and has been translated into several languages. Each section in the scale covers a different domain (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling). Each item is scored on a scale from 0-5 with the first item scored a "0" and representing no disability. The final item is scored a "5" and represents the maximum level of disability. If more than one response in a section is checked, the highest score is chosen. The scores for each section are summed for a final score ranging from 0 to 50. If an item is not answered, the total score is instead calculated as a percentage of the total possible score for all items that were completed.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by pain condition-related medication usage | 6 months
  Pain condition-related medication usage (e.g. opioids, anti-convulsants, anti-depressants, sleep aids, topicals) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by pain condition-related medication usage | 1 Year
  Pain condition-related medication usage (e.g. opioids, anti-convulsants, anti-depressants, sleep aids, topicals) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by pain condition-related medication usage | 2 Years
  Pain condition-related medication usage (e.g. opioids, anti-convulsants, anti-depressants, sleep aids, topicals) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by pain condition-related medication usage | 3 Years
  Pain condition-related medication usage (e.g. opioids, anti-convulsants, anti-depressants, sleep aids, topicals) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by pain condition-related medication usage | 4 Years
  Pain condition-related medication usage (e.g. opioids, anti-convulsants, anti-depressants, sleep aids, topicals) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by pain condition-related medication usage | 5 Years
  Pain condition-related medication usage (e.g. opioids, anti-convulsants, anti-depressants, sleep aids, topicals) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Transcutaneous Oxygen pressure measurement (TcPO2) | 6 months
  Transcutaneous Oxygen pressure measurement (TcPO2) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Transcutaneous Oxygen pressure measurement (TcPO2) | 1 Year
  Transcutaneous Oxygen pressure measurement (TcPO2) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Transcutaneous Oxygen pressure measurement (TcPO2) | 2 Years
  Transcutaneous Oxygen pressure measurement (TcPO2) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Transcutaneous Oxygen pressure measurement (TcPO2) | 3 Years
  Transcutaneous Oxygen pressure measurement (TcPO2) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Transcutaneous Oxygen pressure measurement (TcPO2) | 4 Years
  Transcutaneous Oxygen pressure measurement (TcPO2) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Mean Change in Clinical improvement from baseline to each follow up visit assessed by Transcutaneous Oxygen pressure measurement (TcPO2) | 5 Years
  Transcutaneous Oxygen pressure measurement (TcPO2) will be summarized using mean, standard deviation, median, minimum, maximum, and a 95% confidence interval.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of patient satisfaction | 6 months
  Patient satisfaction will be summarized using counts and percentages
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of patient satisfaction | 1 Year
  Patient satisfaction will be summarized using counts and percentages
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of patient satisfaction | 2 Years
  Patient satisfaction will be summarized using counts and percentages
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of patient satisfaction | 3 Years
  Patient satisfaction will be summarized using counts and percentages
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of patient satisfaction | 4 Years
  Patient satisfaction will be summarized using counts and percentages
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of patient satisfaction | 5 Years
  Patient satisfaction will be summarized using counts and percentages
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of Patient Global Impression of Change (PGIC) for global improvement of the patient. | 6 months
  The PGIC is a categorical rating scale used to evaluate the subject's impression of change in his/her condition since the beginning of the study treatment. The subject will be requested to rate their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale via an interview technique. The categories are as follows: 1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderatly better, 6-better, and 7-a great deal better
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of Patient Global Impression of Change (PGIC) for global improvement of the patient. | 9 months
  The PGIC is a categorical rating scale used to evaluate the subject's impression of change in his/her condition since the beginning of the study treatment. The subject will be requested to rate their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale via telephone calls. The categories are as follows: 1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderatly better, 6-better, and 7-a great deal better
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of Patient Global Impression of Change (PGIC) for global improvement of the patient. | 1 Year
  The PGIC is a categorical rating scale used to evaluate the subject'simpression of change in his/her condition since the beginning of thestudy treatment. The subject will be requested to rate their overallchange in activity limitations, symptoms, emotions and overall qualityof life related to his/her condition on a seven-point categorical scale via an interview technique. The categories are as follows: 1-nochange, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderatly better, 6-better, and 7-a great deal better.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of Patient Global Impression of Change (PGIC) for global improvement of the patient. | 1.5 Year
  The PGIC is a categorical rating scale used to evaluate the subject's impression of change in his/her condition since the beginning of the study treatment. The subject will be requested to rate their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale via telephone calls. The categories are as follows: 1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderatly better, 6-better, and 7-a great deal better
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of Patient Global Impression of Change (PGIC) for global improvement of the patient. | 2 Years
  The PGIC is a categorical rating scale used to evaluate the subject's impression of change in his/her condition since the beginning of the study treatment. The subject will be requested to rate their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale via an interview technique. The categories are as follows: 1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderatly better, 6-better, and 7-a great deal better.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of Patient Global Impression of Change (PGIC) for global improvement of the patient. | 2.5 Years
  The PGIC is a categorical rating scale used to evaluate the subject's impression of change in his/her condition since the beginning of the study treatment. The subject will be requested to rate their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale via telephone calls. The categories are as follows: 1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderatly better, 6-better, and 7-a great deal better
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of Patient Global Impression of Change (PGIC) for global improvement of the patient. | 3 Years
  The PGIC is a categorical rating scale used to evaluate the subject's impression of change in his/her condition since the beginning of the study treatment. The subject will be requested to rate their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale via an interview technique. The categories are as follows: 1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderatly better, 6-better, and 7-a great deal better.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of Patient Global Impression of Change (PGIC) for global improvement of the patient. | 3.5 Years
  The PGIC is a categorical rating scale used to evaluate the subject's impression of change in his/her condition since the beginning of the study treatment. The subject will be requested to rate their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale via telephone calls. The categories are as follows: 1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderatly better, 6-better, and 7-a great deal better
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of Patient Global Impression of Change (PGIC) for global improvement of the patient. | 4 Years
  The PGIC is a categorical rating scale used to evaluate the subject's impression of change in his/her condition since the beginning of the study treatment. The subject will be requested to rate their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale via an interview technique. The categories are as follows: 1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderatly better, 6-better, and 7-a great deal better.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of Patient Global Impression of Change (PGIC) for global improvement of the patient. | 4.5 Years
  The PGIC is a categorical rating scale used to evaluate the subject's impression of change in his/her condition since the beginning of the study treatment. The subject will be requested to rate their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale via telephone calls. The categories are as follows: 1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderatly better, 6-better, and 7-a great deal better
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Rate of Patient Global Impression of Change (PGIC) for global improvement of the patient. | 5 Years
  The PGIC is a categorical rating scale used to evaluate the subject's impression of change in his/her condition since the beginning of the study treatment. The subject will be requested to rate their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale via an interview technique. The categories are as follows: 1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderatly better, 6-better, and 7-a great deal better.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.

CONTACTS AND LOCATIONS:
Overall Officials: Devyani Nanduri, Study Director — Abbott Medical Devices Neuromodulation
Locations (55):
- United States (30):
  - Phoenician Centers for Research & Innovation, Phoenix, Arizona
  - Pain Institute of Southern Arizona, Tucson, Arizona
  - California Orthopedics & Spine, Larkspur, California
  - Restore Orthopedics & Spine Center, Orange, California
  - Foothills Pain Management Clinic, Pomona, California
  - Pacific Research Institute, Santa Rosa, California
  - University of Florida Department of Anesthesia, Gainesville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Goodman Campbell Brain and Spine, Indianapolis, Indiana
  - Nura, Edina, Minnesota
  - Twin Cities Pain Clinic, Edina, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis Pain Consultants, Chesterfield, Missouri
  - Advanced Pain Care, Henderson, Nevada
  - Nevada Advanced Pain Specialists, Reno, Nevada
  - Ainsworth Institute of Pain Management, New York, New York
  - Unity Spine Center, Rochester, New York
  - The Spine & Pain Institute of New York, Staten Island, New York
  - Premier Pain Solutions, Asheville, North Carolina
  - Adena Bone and Joint Center, Chillicothe, Ohio
  - Premier Pain Treatment Institute, Loveland, Ohio
  - Pacific Sports & Spine, Eugene, Oregon
  - Spinal Diagnostics, Tualatin, Oregon
  - Center for Interventional Pain & Spine, Exton, Pennsylvania
  - Expert Pain, Houston, Texas
  - Central Texas Pain Institute, Killeen, Texas
  - Integrated Pain Associates, Killeen, Texas
  - Advanced Pain Care, Round Rock, Texas
  - The Spine & Nerve Center of St Francis Hospital, Charleston, West Virginia
- Australia (2):
  - Metro Pain Group, Clayton, Victoria
  - Precision Brain, Spine & Pain Centre, Kew, Victoria
- Belgium (2):
  - AZ Nikolaas, Sint-Niklaas, Eflndrs
  - AZ Delta vzw, Roeselare, West Flanders
- Germany (9):
  - Universitäts Klinikum Tübingen, Tübingen, Bad-wur
  - Klinikum Ingolstadt GmbH, Ingolstadt, Bavaria
  - Krankenhaus Porz am Rhein, Cologne, Koln
  - Klinikum Duisburg GmbH, Duisburg, N. RHIN
  - Universitaetsklinikum Duesseldorf, Düsseldorf, N. RHIN
  - Krankenhaus Neuwerk Maria von den Aposteln, Mönchengladbach, N. RHIN
  - Kliniken der Stadt Köln-Merheim, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Hospital Gera -Zentrum für interdisziplinäre Schmerztherapie, Gera, Thuringia
- Italy (2):
  - Azienda Ospedaliera Monaldi, Napoli, Campani
  - Fondazione Salvatore Maugeri, Pavia, Lombard
- Netherlands (2):
  - Erasmus MC, Rotterdam, S Holln
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
- Spain (3):
  - Hospital Universitario de Salamanca, Salamanca, Cstleon
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia
- Hôpital du Valais, Sion, Valais, Switzerland
- United Kingdom (4):
  - Norfolk and Norwich Hospital, Norwich, England
  - The Walton Centre, Liverpool, North West England
  - Southmead Hospital, Bristol, Sowest
  - Seacroft Hospital, Leeds, Yorkshire and the Humber

IPD SHARING:
Plan to Share IPD: No